CLINICAL TRIAL: NCT07404813
Title: The Effect of Family Member Voices on Dopamine, Serotonin Levels, and Pain in Patients in Intensive Care Units
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zeliha CENGİZ (Other)
Collaborators: Inonu University (Other)
Responsible Party: Sponsor-Investigator, Zeliha CENGİZ, Associate Professor Dr., Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024/59
Record Dates: First submitted 2026-02-02; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Patient Engagement; Intensive Care (ICU); Family Members' Voices
Keywords: Relatives' Voices; Pain,; serotonin; Dopamine; Satisfaction
MeSH Terms: conditions — Patient Participation; Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: In the experimental group, patients were exposed to a protocol consisting of emotional-content audio recordings obtained from close relatives, each 20 minutes long, with a 10-minute rest between applications, arranged as two sets, and delivered via headphones for a total of 40 minutes. In both groups, behavioral pain assessments were conducted at 0, 20, and 50 minutes, and dopamine and serotonin levels were measured from venous blood samples. To collect study data, a personal information form, Glasgow Coma Scale, Richmond Agitation-Sedation Scale, Behavioral Pain Scale, and a family/patient relative satisfaction questionnaire (FS-ICU-24) were used. For the control group, at 0 minutes 5 mL (5 cc) of venous blood was drawn to measure dopamine and serotonin levels, and behavioral pain scores were recorded. From 0 to 20 minutes, no intervention was performed; however, the patients were exposed to intensive-care unit (ICU) sounds for 20 minutes. A 5 mL venous blood sample was drawn again to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): In the experimental group, patients were exposed to a protocol consisting of emotional-content audio recordings obtained from close relatives, each 20 minutes long, with a 10-minute rest between applications, arranged as two sets, and delivered via headphones for a total of 40 minutes. In the experimental group, behavioral pain assessments were conducted at 0, 20, and 50 minutes, and dopamine and serotonin levels were measured from venous blood samples. To collect study data, a personal information form, Glasgow Coma Scale, Richmond Agitation-Sedation Scale, Behavioral Pain Scale, and the FS-ICU-24 patient/family satisfaction questionnaire were used.
  Interventions: Other: Experimental Group
- control group (No Intervention): In this group, no intervention is performed, and the patients are exposed to ICU sounds. For the control group, at 0 minutes 5 mL (5 cc) of venous blood was drawn to measure dopamine and serotonin levels, and behavioral pain scores were recorded. From 0 to 20 minutes, no intervention was performed; however, the patients were exposed to intensive-care unit (ICU) sounds for 20 minutes. A 5 mL venous blood sample was drawn again to check dopamine and serotonin levels, and behavioral pain scores were recorded. The patients were then exposed to normal ICU sounds for 10 additional minutes. From 30 to 50 minutes, again without any intervention, patients were exposed to ICU sounds for 20 minutes; a 5 mL venous blood sample was drawn to measure dopamine and serotonin levels, and behavioral pain scores were recorded.

INTERVENTIONS:
Other: Experimental Group — The patients' relatives were given a detailed explanation of the procedures and were asked to fill out a patient/family satisfaction questionnaire. The topics to be discussed by the patient's family members were defined within a framework, and audio recordings were obtained. At 0 minutes, 5 mL of venous blood was drawn to assess dopamine and serotonin levels, and behavioral pain scores were recorded. Between 0 and 20 minutes, for 20 minutes, the audio recordings were played to the patient via headphones, 5 mL of venous blood was drawn again to assess dopamine and serotonin levels, and behavioral pain scores were recorded. At 10 minutes, the headphones were removed and the patient was exposed to normal ICU sounds. Between 30 and 50 minutes, again for 20 minutes, the audio recordings were played to the patient via headphones, 5 mL of venous blood was drawn again to assess dopamine and serotonin levels, and behavioral pain scores were recorded.
  Arms: experimental group

SUMMARY:
In intensive care units, the frequent use of analgesics leads to polypharmacy and increased costs for patients. By embracing a patient-centered care principle, nursing believes that patients may be happier and experience reduced pain when they hear the voices of their familiar ones, thereby directly improving their quality of life. Listening to the voices of family members is expected to have positive effects on patients due to its ease of implementation, low cost, and non-invasive nature.

DETAILED DESCRIPTION:
In intensive care units, the frequent use of analgesics leads to excessive medication use and increased costs for patients. By embracing a patient-centered care principle, nursing believes that patients may be happier and experience reduced pain when they hear the voices of their familiar ones, thereby directly improving their quality of life. Listening to the voices of family members is expected to have positive effects on patients due to its ease of implementation, low cost, and non-invasive nature. This study was planned to be conducted between 01.03.2025 and 01.03.2026 at İnönü University Turgut Özal Medical Center General Surgery Intensive Care, Neurology Intensive Care, and Neurosurgery Intensive Care units. The aim was to determine the effects of family members' voices on dopamine and serotonin levels and pain in ICU patients, as well as family members' satisfaction levels. The study was designed as a randomized controlled trial. The sample for the study would consist of 78 ICU patients (experimental group = 39, control group = 39) treated in these clinics, determined by power analysis for the data collection dates. In the experimental group, recordings of emotionally charged voices from family members were played to patients using headphones for a total of 40 minutes, structured as 2 sets of 20 minutes each with a 10-minute rest between applications. In both groups, behavioral pain assessment was planned at 0, 20, and 50 minutes, and dopamine and serotonin levels would be measured from venous blood samples. To collect study data, a Personal Information Form, Glasgow Coma Scale, Richmond Agitation-Sedation Scale, Behavioral Pain Scale, and a family member satisfaction questionnaire (FS-ICU-24) were used. Power analysis conducted with the G*Power program considered an effect size of 0.20, a significance level of 0.05, a 95% confidence interval, and 0.95 power.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 and 65 years old.
* Must be admitted to an intensive care unit (ICU).
* Must not have been fed in the last hour.
* Glasgow Coma Scale (GCS) score between 3 and 8.
* To agitation in deep coma, the Richmond Agitation-Sedation Scale (RASS) score must be between -3 and +2.

Exclusion Criteria:

* Having a known hearing-related illness or having undergone a surgical procedure involving the ear.
* Having taken any of the hormones cortisol, serotonin, or dopamine within the last 48 hours.
* Having taken any analgesic within the last 4 hours.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Compared with Baseline, at 20 And 50 Minutes after The Patient-Family Voice Recordings Were Played, Dopamine and Serotonin Levels İncreased and Pain Decreased According to The Behavioral Pain Scale. | Changes in dopamine, serotonin, and pain at 0, 20, and 50 minutes after the patient's family voices were played.
  An increase in dopamine and serotonin levels in the venous blood of patients compared with the control group, and a low score on the measured Behavioral Pain Scale relative to baseline (with 10 being the highest and 1 the lowest), would indicate that the audio recordings are a positive intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Malatya Turgut Ozal Medical Center, Malatya, Malatya
  - Şırnak Üniversitesi, Şırnak, Merkez

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yu WC, Chiang MC, Lin KC, Chang CC, Lin KH, Chen CW. Effects of maternal voice on pain and mother-Infant bonding in premature infants in Taiwan: A randomized controlled trial. J Pediatr Nurs. 2022 Mar-Apr;63:e136-e142. doi: 10.1016/j.pedn.2021.09.022. Epub 2021 Sep 30. PMID 34602338
- [Result] Tıbık, R., & Şener, D. K. (2024). Preterm Yenidoğanlara Orogastrik Tüp Takma İşlemi Sırasında Dinletilen Anne Sesi ve Beyaz Gürültünün Ağrı Düzeyi ve Fizyolojik Parametrelere Etkisi: Randomize Kontrollü Çalışma. Bandırma Onyedi Eylül Üniversitesi Sağlık Bilimleri ve Araştırmaları Dergisi, 6(1), 109-119.
- See also: Tıbık, R. ve Şener, DK (2024). Preterm Yenidoğanlara Orogastrik Tüp Takma İşlemi Sırasında Dinletilen Anne Sesi ve Beyaz yağının Ağrı Düzeyi ve Fizyolojik Parametrelere Etkisi: Rastgele Kontrollü Çalışma. — https://dergipark.org.tr/en/pub/boneyusbad/article/1406650